CLINICAL TRIAL: NCT02150070
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Intravenous Administration of ASP2408 Manufactured From a New Production Clone and Following Single Ascending Doses of Subcutaneous Injections in Healthy Subjects
Brief Title: A Study to Evaluate a Single Intravenous (IV) Dose Using a New Manufactured Clone and Single Ascending Doses of Subcutaneous (SC) Injections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2408-CL-0102
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Pharmacokinetics of ASP2408; Healthy Subjects
Keywords: Healthy subjects; ASP2408; Rheumatoid arthritis; Safety and Tolerability; Pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ASP2408

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Intravenous ASP2408 (Experimental)
  Interventions: Drug: ASP2408
- Subcutaneous ASP2408 low dose (Experimental)
  Interventions: Drug: ASP2408
- Subcutaneous ASP2408 middle dose (Experimental)
  Interventions: Drug: ASP2408
- Subcutaneous ASP2408 high dose (Experimental)
  Interventions: Drug: ASP2408
- Intravenous Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Subcutaneous Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2408 — Intravenous (IV) infusion and subcutaneous (SC) injection
  Arms: Intravenous ASP2408; Subcutaneous ASP2408 high dose; Subcutaneous ASP2408 low dose; Subcutaneous ASP2408 middle dose
Drug: Placebo — Intravenous (IV) infusion and Subcutaneous (SC) injection
  Arms: Intravenous Placebo; Subcutaneous Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics (PK) after intravenous (IV) administration of ASP2408 manufactured from a new production clone and also following single ascending doses of subcutaneous (SC) injections of the same clinical trial material.

DETAILED DESCRIPTION:
The four doses will be studied in sequential cohorts of 8 subjects each, starting with the IV dose, followed by the subcutaneous doses in ascending order of dose. Within each cohort, subjects will be randomized to either active drug or matching placebo in a 3:1 ratio (6 active and 2 placebo).

All subjects in each arm will be confined for 8 days and followed for a minimum of 90 days up to 9 months if necessary. Subjects who have study drug terminated should remain in the study, if possible and have scheduled procedures and follow-up.

Subjects who have detectable blood levels of ASP2408 after Day 90 will be unblinded and followed monthly until ASP2408 levels are below the limit of quantification. In addition, subjects who have persistent anti-ASP2408 antibodies after Day 90 will be unblinded and followed every 30 (± 3) days for up to 9 months until the level of these antibodies are declining, no longer detectable, and/or have no clinical consequence.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, a maximum of 92.5 kg and has a body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* The subject's 12-lead electrocardiogram (ECG) results are normal
* The female subject must be at least two years postmenopausal OR surgically sterile and not pregnant or lactating
* The male subject agrees to the use of male condoms until the end of study or 60 days post dose, whichever is longer

Exclusion Criteria:

* The subject has a history of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy excluding adequately-treated non-melanoma skin cancer
* The subject has a history of severe allergic or anaphylactic reactions
* The subject is a female of childbearing potential
* The subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within the past 2 years (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* The subject has a positive test for alcohol or drugs of abuse
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check-in
* The subject has a past history of opportunistic infection
* The subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or mean pulse rate higher than 100 beats per minute (bpm)
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive tuberculosis (TB) skin test, Quantiferon Gold test or T-SPOT® test
* The subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody
* Subject's alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values are greater than 1.5 times the upper limit of normal
* Subject's laboratory test results are outside the normal limits and considered to be clinically significant
* The subject received any vaccine within 60 days prior to study drug administration
* The subject received any systemic immunosuppressant agent within 2 months prior to study drug administration
* The subject has previously received any antibody or therapeutic biologic product prior to study drug administration
* The subject received any systemic steroid within 2 months or steroid inhaler within 1 month prior to study drug administration
* The subject has had treatment with prescription, non-prescription or complementary and alternative medicines (CAM) within 14 days prior to study drug administration with the exception of stable hormone replacement therapy (HRT) and/or intermittent acetaminophen (to a maximum of 2 g/day)
* The subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* The subject is participating in another clinical trial or has participated in another dose group of the current trial
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* The subject has any other condition which precludes the subject's participation in the trial
* The subject has a history of heavy smoking or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP2408: AUClast | Days 1-9, 11, 13, 15, 22, 29, 43, 60, and 90
  Area under the concentration - Time curve from time 0 up to the last quantifiable concentration (AUClast)
Pharmacokinetic parameter of ASP2408: AUCinf | Days 1-9, 11, 13, 15, 22, 29, 43, 60, and 90
  Area under the concentration - Time curve from time 0 extrapolated to infinity (AUCinf)
Pharmacokinetic parameter of ASP2408: Cmax | Days 1-9, 11, 13, 15, 22, 29, 43, 60, and 90
  Maximum concentration (Cmax)
Safety assessed by adverse events (AEs), laboratory tests, immunoglobulin quantification (class), 12-lead electrocardiograms, vital signs and anti-ASP2408 antibody formation | Up to day 90

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP2408: tmax, t 1/2, Vz/F, CL/F and F (%) | Days 1-9, 11, 13, 15, 22, 29, 43, 60, and 90
  Time to attain Cmax (tmax), apparent terminal elimination half-life (t 1/2), apparent volume of distribution (Vz/F), apparent body clearance (CL/F) and absolute bioavailability (F%)
Pharmacodynamic Profile: CD80 and CD86 receptor occupancy, peripheral lymphocyte subset quantification (leukocyte phenotypes) and total lymphocyte count | Days 1-3, 5, 8, 15, 22, 29, 43, 60 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel International, Baltimore, Maryland, United States